CLINICAL TRIAL: NCT01670942
Title: The Effects of Hypobaric Conditions on Small, Traumatic Pneumothoraces
Brief Title: Hypobaria and Traumatic Pneumothorax
Status: Completed | Type: Observational
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Principal Investigator, Sarah Majercik, MD, MBA, FACS, Intermountain Health Care, Inc.
Other Study IDs: IRB#1024157
Record Dates: First submitted 2012-08-18; First posted 2012-08-23 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Pneumothorax
Keywords: pneumothorax; trauma; commercial air travel
MeSH Terms: conditions — Pneumothorax; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Traumatic Pneumothorax1: hypobaric chamber
  Interventions: Other: hypobaric chamber

INTERVENTIONS:
Other: hypobaric chamber — We will use a large (26 tons) multi-place hyperbaric and hypobaric chamber at IMC in Murray, Utah (elevation 1500m or 4500ft, average ambient barometric pressure 645mm Hg). In the hypobaric study, the barometric pressure will be lowered to 554mm Hg (phase 1) or 471mm Hg (phase 2) over 20 minutes and held there for two hours.

SUMMARY:
The purpose of this research is to see if people who have had a collapsed lung that has been re-expanded can be safely taken to an elevation that a person might experience while in a commercial airplane without having their lung partially collapse again, or have any symptoms such as feeling short of breath or having oxygen levels in the blood decrease while at the simulated altitude.

The investigators hypothesize that subjects who have had a collapsed lung that has been re-expanded will not have any adverse symptoms or signs while subjected to a simulated altitude of 8400 feet (565mm Hg) or 12650 ft (471mm Hg).

DETAILED DESCRIPTION:
The investigators will study patients who have been diagnosed with a unilateral traumatic pneumothorax that has been treated. Treatment for pneumothorax may consist of high-flow oxygen therapy in the case of very small or "occult" pneumothorax, or tube thoracostomy ("chest tube") in the case of larger pneumothorax. Treatment for pneumothorax will be at the discretion of the attending trauma surgeon. Once the pneumothorax has radiographically resolved, the chest tube, if used, has been removed, and prior to discharge from the hospital, subjects will undergo a two hour stay in a hypobaric chamber. In the first phase of the study, they will undergo a two hour stay in a hypobaric chamber at a barometric pressure of 565mm Hg, simulating the change in pressure from Salt Lake City to a cruising airliner. If subjects in the first phase do not suffer any adverse events, the investigators will proceed with the second phase. In the second phase of the study, subjects will undergo a two hour stay in the hypobaric chamber at a barometric pressure of 471mm Hg, simulating the change in pressure from sea level to a cruising airliner. Prior to the hypobaric exposure, and at the conclusion of the two hours under hypobaric conditions, single view chest radiographs will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Inpatient status on trauma surgery service
2. An established diagnosis of pneumothorax with a traumatic etiology (patients with iatrogenic pneumothorax from attempted central venous line placement will be considered to have a traumatic etiology)
3. Age ≥ 18 at the time of injury

Exclusion Criteria:

1. Pregnancy
2. Unable to give informed consent
3. Pneumothorax which does not satisfactorily resolve after treatment with tube thoracostomy and requires operative intervention such as video assisted thoracoscopic surgery (VATS) or thoracotomy
4. Pneumothorax requiring tube thoracostomy where the tube has been removed for < 4 or > 48 hours
5. Head injury with GCS < 15 at time of evaluation for study
6. Other injuries or conditions which would preclude participant's ability to remain in chamber for two hours
7. NYHA class III or IV heart failure, active coronary artery disease, arrhythmias, pacemakers, implantable cardiac defibrillator, pulmonary hypertension, claustrophobia
8. Severe obstructive or restrictive lung disease
9. Chronic hypoxemia requiring supplemental oxygen
10. Hypoxemia for any reason (pulmonary contusion, atelectasis, pneumonia, etc.) requiring > 3 liters supplemental oxygen at the time of entry into the study
11. Inability to tolerate the confines of the chamber

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with unilateral pneumothorax of traumatic etiology that has been treated with oxygen, observation, or tube thoracostomy
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in pneumothorax size | baseline and 2 hours
  Will document pneumothorax size before simulated altitude, and size after being at simulated altitude for two hours

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Majercik, MD, MBA, Principal Investigator — Intermountain Health Care, Inc.; Lindell Weaver, MD, Study Director — Intermountain Health Care, Inc.
Locations (1):
- Intermountain Medical Center, Murray, Utah, United States